CLINICAL TRIAL: NCT04758325
Title: A Prospective Registry Study on Biological Disease Profile, Intervention Type and Clinical Outcome in Adolescent and Adult Patients With Soft-tissue and Bone Sarcoma
Brief Title: The Sarcoma Biology and Outcome Project
Acronym: SarcBOP
Status: Recruiting | Type: Observational
Sponsor: Prof. Dr. Richard F Schlenk (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Richard F Schlenk, Head of NCT trials center and Clinical Trials, University Hospital Heidelberg
Organization: University Hospital Heidelberg (Other)
Other Study IDs: TMO1902
Record Dates: First submitted 2021-02-04; First posted 2021-02-17 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Sarcoma; Malignant Mesenchymoma; Sarcoma of Bone and Connective Tissue
Keywords: rare disease; database; treatment; research; molecular diagnostic; translational approach; interdisciplinary approach
MeSH Terms: conditions — Sarcoma; Malignant mesenchymal tumor; Osteosarcoma; Rare Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
SarcBOP - An interdisciplinary and translational registry

SarcBOP aims to establish a database that integrates every aspect possibly relevant to sarcoma treatment and research. SarcBOP thus will not be limited to specific questions or patient groups, but instead will build a comprehensive database including clinical, pathologic, and radiologic information, multi-layered molecular data, and patient-reported outcomes, combined with a dedicated biobank for tissue samples and liquid biopsies. As the study integrates seamlessly with the clinical activities of the Heidelberg Sarcoma Center, the Molecular Diagnostics Program of NCT Heidelberg, including the NCT/DKTK MASTER Program, and with the NCT Trial Center, including the PMO Clinical Trials Program, SarcBOP will generate a comprehensive and continuously growing resource for clinicians, researchers, and, finally, patients.

DETAILED DESCRIPTION:
The following data are collected and stored:

* Demographics
* Comorbidities
* Clinical characteristics at diagnosis, relapse and progression
* Radiologic images
* Histological images
* Treatments including DRG and OPS data, including detailed information on surgical, radiation, and medical therapy as well as treatment relevant follow-up data
* Longitudinal disease assessments
* Clinical outcome
* Genomic, transcriptomic, epigenomic and proteomic data
* Patient reported outcomes

Furthermore, biological samples are collected and processed by the Sample Processing Laboratory of the Heidelberg Center for Personalized Oncology and the NCT Biobank.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or proven diagnosis of soft-tissue or bone sarcoma (STBS)
* Age ≥12 years
* Ability to understand nature and individual consequences of the registry
* Written informed consent
* Subjects who are physically or mentally capable of giving consent

Exclusion Criteria:

• Severe neurological or psychiatric disorder interfering with the ability to give written informed consent

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Soft-tissue and Bone Sarcoma
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-07-23 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5 years
  The length of time from the date of diagnosis disease, that patients diagnosed with are still alive
overall survival | 10 years
  The length of time from the date of diagnosis disease, that patients diagnosed

SECONDARY OUTCOMES:
progression free survival | 5 years
  length of time during and after treatment, that a Patient lives with the disease without getting worse

OTHER OUTCOMES:
Core questionnaire QLQ-C30 | 5 years
  Standardized Quality of Life Assessment, Higher values are better
Fatigue module QLQ-FA12 | 5 years
  Standardized Quality of Fatigue, Higher values are worse
PHQ-4 (anxiety and depression) | 5 years
  Standardized Quality of anxiety and depression, Higher values are worse
FACT-cog (cognitive function) | 5 years
  Standardized Quality of cognitive function, Higher values are better
DASH | 5 years
  Disability of the arm, shoulder and hand, lower values are better
EFAS | 5 years
  European foot and ankle society, higher values are better
OKS | 5 years
  Oxford knee score function and pain questionnaire after total knee replacement surgery, (TKR), higher values are better
MSTS | 5 Years
  Musculoskeletal tumor society score, higher values are better
ODI | 5 Years
  Oswestry back pain disability questionnaire after spinal surgery, lower values are better
OHS | 5 years
  Oxford hip score - Function and pain questionnaire after hip replacement surgery, higher values are better
PSQI | 5 years
  Pittsburgh Sleep Quality Index, Higher values are worse
Sociodemographics | Baseline only
  Sociodemographic data

CONTACTS AND LOCATIONS:
Overall Officials: Richard F. Schlenk, Prof.Dr.med, Principal Investigator — National Center for Tumour Disease; Christoph E. Heilig, Dr. med., Study Director — National Center for Tumour Disease; Stefan Fröhling, Prof. Dr., Study Director — National Center for Tumour Disease
Locations (1):
- National Center for Tumour Diseases, University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: official website of SarcBOP — http://www.nct-heidelberg.de/sarcbop